CLINICAL TRIAL: NCT03885414
Title: Virtual Reality Exposure Therapy for Public Speaking Anxiety: A Multiple-baseline Effectiveness Trial
Brief Title: Virtual Reality Exposure Therapy for Public Speaking Anxiety
Acronym: VRETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: PBM (Unknown); Mimerse (Unknown)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRETA
Record Dates: First submitted 2019-03-11; First posted 2019-03-21 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Public Speaking; Social Anxiety; Social Anxiety Disorder, Performance Only
MeSH Terms: conditions — Speech; Phobia, Social | interventions — Virtual Reality Exposure Therapy; Implosive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Multiple baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OST-VRET + in-vivo transition program (Experimental): One-session treatment (OST) VRET on-location with clinical psychologist (3 hours), followed by a therapist-guided, four-week online program encouraging transition to real-world, in-vivo exposure exercises.
  Interventions: Behavioral: In-session Virtual Reality exposure therapy; Behavioral: Internet-administered transition program

INTERVENTIONS:
Behavioral: In-session Virtual Reality exposure therapy — A series of exposure exercises (speech exercises) in front of a virtual audience, focusing on promoting inhibitory learning, with audio-feedback.
  Other Names: Virtual reality therapy; Exposure therapy; Cognitive behavioral therapy
Behavioral: Internet-administered transition program — Four-module internet program with weekly therapist guidance, focusing on transitioning to in-vivo exposure in everyday settings.
  Other Names: Internet intervention

SUMMARY:
Virtual Reality exposure therapy (VRET) is an efficacious treatment for anxiety disorders but has yet to be implemented in regular care settings. This is arguably due to the limitations of the past generation of VR technology, which was expensive, inaccessible, cumbersome and hard to use. With the advent of consumer VR technology, VRET is now ready for implementation in regular care. This multiple-baseline trial will examine the effectiveness of VRET for public speaking anxiety (PSA) when delivered under real-world conditions at an ordinary, non-specialized mental health clinic, by clinical psychologist with only brief VRET training. Participants will either be self-referred specifically for this treatment, or come through ordinary clinical channels. Self-rated PSA will serve as primary outcome measure and will be measured three times prior to treatment (at screening and twice after a diagnostic screening telephone interview) , four times after onset, at the end of the treatment period, and three months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have substantial public speaking anxiety (PSAS >= 60)
* Can travel to PBM clinic on one occasion and pay stipulated patient fee
* Can speak and understand sufficient Swedish
* Have stable access to the internet

Exclusion Criteria:

* Deficits in sight or balance impacting the VR-experience
* A severe psychiatric disorder better treated elsewhere, including current major depression, alcohol or drug abuse, bipolarity, psychosis or similar
* Active psychopharmacological treatment, unless stable for last 3 months
* Other ongoing psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline: Public Speaking Anxiety Scale | Change from baseline: (1) five days after interview, (2) ten days after interview, (3) 7 days post-OST, (4) 14 days post-OST (5) 21 days post-OST (6) 28 days post-OST, (7) 35 days post-OST, (8) 125 days post-PST
  Canonical total score will be used. Measure is self-rated, online. Swedish translation of the original PSAS (Bartholomay & Houlihan, 2016)

SECONDARY OUTCOMES:
Change from baseline: Brunnsviken Brief Quality of life scale | Change from baseline: (1) 7 days post-OST, (4) 35 days post-OST, (5) 125 days post-PST
  Canonical total score will be used. Measure is self-rated, online.
Change from baseline: Liebowitz Social Anxiety Scale Self-Report | Change from baseline: (1) 7 days post-OST, (2) 35 days post-OST, (3) 125 days post-PST
  Canonical total score will be used. Measure is self-rated, online.
Change from baseline: Brief Fear of Negative Evaluation Scale | Change from baseline: (1) 7 days post-OST, (2) 35 days post-OST, (3) 125 days post-PST
  Canonical total score will be used. Measure is self-rated, online.
Change from baseline: Patient Health Questionnaire 9-item | Change from baseline: (1) 7 days post-OST, (2) 35 days post-OST, (3) 125 days post-PST
  Canonical total score will be used. Measure is self-rated, online.
Change from baseline: Generalized Anxiety Disorder 7-item | Change from baseline: (1) 7 days post-OST, (2) 35 days post-OST, (3) 125 days post-PST
  Canonical total score will be used. Measure is self-rated, online.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, PhD, Principal Investigator — Stockholm University
Locations (1):
- Department of Psychology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous outcome measure IPD will be made available upon request from academic researchers.

REFERENCES:
- [Background] Lindner P, Miloff A, Fagernas S, Andersen J, Sigeman M, Andersson G, Furmark T, Carlbring P. Therapist-led and self-led one-session virtual reality exposure therapy for public speaking anxiety with consumer hardware and software: A randomized controlled trial. J Anxiety Disord. 2019 Jan;61:45-54. doi: 10.1016/j.janxdis.2018.07.003. Epub 2018 Jul 24. PMID 30054173
- See also: Study website (Swedish) — https://www.iterapi.se/sites/vreta/